CLINICAL TRIAL: NCT03901690
Title: Betaglucin 0.2% Gel Versus Imiquimod Cream 5% in the Treatment of Anogenital Warts in 102 Individuals Older Than 18 Years.
Brief Title: Betaglucin 0.2% Versus Imiquimod 5% in Treatment of Ano-genital Warts: Combined Results From Triple Blind Controlled Study
Acronym: BETAGENWART
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro de Investigaciones Medicas y Ensayos Clinicos Dr Italo Fabbri (Network)
Collaborators: CALOX Laboratories (Unknown); Bioanalisis (Unknown)
Responsible Party: Principal Investigator, Alejandro Pérez Fabbri MD FACOG, Doctor in Medicine. Executive Director CIMIF, Centro de Investigaciones Medicas y Ensayos Clinicos Dr Italo Fabbri
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-001
Record Dates: First submitted 2019-03-28; First posted 2019-04-03 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Genital Wart Virus Infection
Keywords: Betaglucin soluble gel; Ano-genital warts; Clearance; Human papillomavirus
MeSH Terms: interventions — Imiquimod

STUDY DESIGN:
Intervention Model Description: prospective triple-blind randomized controlled clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In this clinical trial, the masking is triple because neither the participants nor the researchers nor the outcomes assessor will know exactly which drug will receive.
  Only through a list created mathematically by Prof R Fentin will serve as a unique guide for the administration masked either beta-glucan gel or imiquimod in cream. Both packaged in the same tube without labeling on the outside.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm Betaglucin (Experimental): It will be composed of 51 individuals between 18 and 50 years old with anogenital warts to which will be applied betaglucin gel at 0.2%.
  Interventions: Drug: Betaglucin soluble gel 0.2%
- Arm Imiquimod (Active Comparator): 51 individuals between the ages of 18 and 50 will receive 5% imiquimod.
  Interventions: Drug: Imiquimod 5% cream

INTERVENTIONS:
Drug: Betaglucin soluble gel 0.2% — With the prior informed consent of the 51 study participants, 5 grams of 0.2% soluble betaglucin gel will be self-applied every 12 hours for 5 days. Both groups will receive an unlabeled tube so that none of the study participants will know what topical treatments they are receiving.
  Arms: Arm Betaglucin
Drug: Imiquimod 5% cream — With the prior informed consent of the 51 study participants, 1 gram of 5% imiquimod will be self-applied once a day for 5 days. Both groups will receive an unlabeled tube so that neither study participant knows what topical treatments they are receiving.
  Arms: Arm Imiquimod

SUMMARY:
In order to determine the Efficacy of Betaglucin 0.2% in gel vs Imiquimod 5% cream in the treatment of 102 individuals older than 18 years with anogenital warts trials in two arms 51 with Betaglucin 0.2% and 51 with Imiquimod 5%.

DETAILED DESCRIPTION:
Betaglucin soluble gel at 0.2% is produced in Costa Rica by a biochemical researcher. Obtained by chemical process improves the immune response by increasing 80 times the number of macrophages and Natural Killer cells. Specifically in human papillomavirus-related anogenital warts.

As clinical researchers, the investigators pretend to determine the therapeutic efficacy of betaglucin 0.2 % gel compared with Imiquimod 5% cream in two groups of individuals from 18 to 50 years old males and females.

Based in mathematics and biostatistics formula used by Professor Roman Fentin, French academic working in the University of Costa Rica. Medicine Faculty in San Jose the number of participants should be 102.

Divided into two arms. Arm betaglucin 0.2% 51 individuals treated with betaglucin soluble gel at 0.2% Arm imiquimod 5% 51 individuals treated with imiquimod cream at 5 % After three months of follow-up of all individuals, will be classified as clearance, partially cured and not cured.

The plan of analysis will be:

* Chi-square test between the two groups (depending on the treatment) and the success or not of the treatment.
* Logistic model with a dependent variable the success or not of the treatment and with independent variables the treatment, sex, age. It will make it possible to verify that the differences observed in 1 are not due to another factor.
* Logistic model with a dependent variable the success or not of the treatment and with independent variables the treatment, the sex, the age, and an interaction sex-age. It will allow us to observe if there is a difference in the result according to the patient's sex.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 50 years with anogenital wart visible on physical examination and positive for HPV 6 and 11 by polymerase chain reaction (PCR) test with detection by agarose gel electrophoresis.

Exclusion Criteria:

* Pregnant women.
* Vaccinated against human papillomavirus (Gardasil, Gardasil 9 or Cervarix).
* Patients Immunosuppressed by drugs (Chemotherapy, Corticoids, use of antibiotics for more than 7 days and/or antituberculous treatment.)
* Molluscum contagiosum.
* Skin Appendages.
* Urethral prolapse.
* Botryoid sarcoma.
* Herpes type II.
* History of anogenital surgery in the last 4 weeks.
* Intake of natural products or immunomodulators.
* Patients who have received 5% imiquimod cream.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2019-08-27 (Actual); Primary Completion 2020-03-10 (Estimated); Study Completion 2020-05-20 (Estimated)

PRIMARY OUTCOMES:
Cure Rate | 3 months
  Completely cured will be those that present a disappearance of 80% or more of the initial volume of the wart, partially cured will be a decrease of at least 50%-79% of the initial volume of the lesion using a measurement rule applied to the larger diameter of this and not cured those that present a reduction of less than 50% of the initial volume.

CONTACTS AND LOCATIONS:
Overall Officials: Romain Fantin, PhD. Math, Study Chair — Centro de Investigaciones Medicas y Ensayos Clinicos Dr Italo Fabbri
Locations (1):
- Clínica San Dominic, Managua, Nicaragua

IPD SHARING:
Plan to Share IPD: Yes
There is a timeline that includes a start date, end date, informed consent signature, study protocol, statistical analysis plan, informed consent form, clinical study report.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Available on May 2019 until May 2021
Access Criteria: Available for clinical researchers, professors and health care providers
URL: http://cimif.org

REFERENCES:
- [Background] Baker DA, Ferris DG, Martens MG, Fife KH, Tyring SK, Edwards L, Nelson A, Ault K, Trofatter KF, Liu T, Levy S, Wu J. Imiquimod 3.75% cream applied daily to treat anogenital warts: combined results from women in two randomized, placebo-controlled studies. Infect Dis Obstet Gynecol. 2011;2011:806105. doi: 10.1155/2011/806105. Epub 2011 Aug 24. PMID 21876641
- [Result] Scardamaglia P, Carraro C, Mancino P, Stentella P. [Effectiveness of the treatment with beta-glucan in the HPV-CIN 1 lesions]. Minerva Ginecol. 2010 Oct;62(5):389-93. Italian. PMID 20938424